CLINICAL TRIAL: NCT00256152
Title: Asymptomatic Atrial Fibrillation and Stroke Evaluation in Pacemaker Patients and the Atrial Fibrillation Reduction Atrial Pacing Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRD291
Record Dates: First submitted 2005-09-10; First posted 2005-11-21 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Hypertension; Atrial Fibrillation
Keywords: Atrial fibrillation; Pacemaker; AF suppression pacing; Indications for Pacemaker Implantation due to sinus node or atrio-ventricular node disease
MeSH Terms: conditions — Hypertension; Atrial Fibrillation

ARMS (2):
- AF Suppression OFF (No Intervention)
- AF Suppression ON (Experimental)
  Interventions: Device: AF Suppression Pacing Algorithm

INTERVENTIONS:
Device: AF Suppression Pacing Algorithm
  Arms: AF Suppression ON

SUMMARY:
In patients with a standard indication for pacing and no previous history of AF, detection of Atrial High Rate Episodes predicts an increased risk of stroke and systemic embolism.

Overdrive atrial pacing with the AF Suppression algorithm will reduce the risk of symptomatic AF in patients with standard indication for pacing and no previous history of AF.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 65 years
2. History of hypertension requiring pharmacological therapy (≥ 4 weeks of therapy).
3. Recent (< 8 weeks) St. Jude Medical Inc. pacemaker implant (IDENTITY® Adx DR (Model 5386/5380)), ICD implant (EPIC 2 or Atlas 2) or other St. Jude Medical Inc. pacemaker or ICD with the same capabilities.
4. In pacemaker patients only the primary indication for pacing is sinus or AV node disease.

Exclusion Criteria

1. Previous documented AF, atrial flutter (lasting greater than 5 minutes), or other sustained SVT (not including episodes detected by the device)
2. Geographic/social or psychiatric factor likely to interfere with follow-up
3. Requirement for oral anticoagulation (heart valve, deep vein thrombosis, etc.)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2580 (Actual)
Dates: Start 2004-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Composite of ischemic stroke & Non-CNS systemic embolism | 3 years
Symptomatic or Asymptomatic AT documented by ECG | 3 years

SECONDARY OUTCOMES:
Myocardial infarction [MI], Vascular death Composite of stroke, MI or vascular death | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Connolly, MD, Study Chair — McMaster University; Stephan Hohnloser, MD, Study Chair — Goethe University; Carlos Morillo, MD, Principal Investigator — McMaster University; Jeff Healey, MD, Principal Investigator — McMaster University; Carsten Israel, MD, Principal Investigator — Goethe University; Michael Gold, MD, Principal Investigator — Medical University of South Carolina; Chu-Pak Lau, MD, Principal Investigator — The University of Hong Kong; Alessandro Capucci, MD, Principal Investigator — Ospedale Clinic, Piacenza Italy
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Benz AP, Wang J, McIntyre WF, Wong JA, Crystal E, Shurrab M, Israel CW, Hohnloser SH, Gold MR, Connolly SJ, Healey JS. Active-Fixation Atrial Leads and the Risk of Atrial Fibrillation: Insights From ASSERT. Circ Arrhythm Electrophysiol. 2020 Sep;13(9):e008655. doi: 10.1161/CIRCEP.120.008655. Epub 2020 Jul 23. No abstract available. PMID 32701364
- [Derived] Perera KS, Sharma M, Connolly SJ, Wang J, Gold MR, Hohnloser SH, Lau CP, Van Gelder IC, Morillo C, Capucci A, Israel CW, Botto G, Healey JS. Stroke type and severity in patients with subclinical atrial fibrillation: An analysis from the Asymptomatic Atrial Fibrillation and Stroke Evaluation in Pacemaker Patients and the Atrial Fibrillation Reduction Atrial Pacing Trial (ASSERT). Am Heart J. 2018 Jul;201:160-163. doi: 10.1016/j.ahj.2018.03.027. Epub 2018 Apr 18. PMID 29764671
- [Derived] Brambatti M, Connolly SJ, Gold MR, Morillo CA, Capucci A, Muto C, Lau CP, Van Gelder IC, Hohnloser SH, Carlson M, Fain E, Nakamya J, Mairesse GH, Halytska M, Deng WQ, Israel CW, Healey JS; ASSERT Investigators. Temporal relationship between subclinical atrial fibrillation and embolic events. Circulation. 2014 May 27;129(21):2094-9. doi: 10.1161/CIRCULATIONAHA.113.007825. Epub 2014 Mar 14. PMID 24633881
- [Derived] Lau CP, Gbadebo TD, Connolly SJ, Van Gelder IC, Capucci A, Gold MR, Israel CW, Morillo CA, Siu CW, Abe H, Carlson M, Tse HF, Hohnloser SH, Healey JS; ASSERT investigators. Ethnic differences in atrial fibrillation identified using implanted cardiac devices. J Cardiovasc Electrophysiol. 2013 Apr;24(4):381-7. doi: 10.1111/jce.12066. Epub 2013 Jan 28. PMID 23356818
- [Derived] Hohnloser SH, Healey JS, Gold MR, Israel CW, Yang S, van Gelder I, Capucci A, Lau CP, Fain E, Morillo CA, Ha A, Carlson M, Connolly SJ; ASSERT Investigators. Atrial overdrive pacing to prevent atrial fibrillation: insights from ASSERT. Heart Rhythm. 2012 Oct;9(10):1667-73. doi: 10.1016/j.hrthm.2012.06.012. Epub 2012 Jun 12. PMID 22698765
- [Derived] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222